CLINICAL TRIAL: NCT06041945
Title: Saving by Artificial Intelligence for Virtual Endoscopy Biopsy Artificial Intelligence to Implement Cost-saving Strategies for Colonoscopy Screening Based on in Vivo Prediction of Polyp Histology
Brief Title: Artificial Intelligence to Implement Cost-saving Strategies for Colonoscopy Screening Based on in Vivo Prediction of Polyp Histology
Acronym: SAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3483 - SAVE
Record Dates: First submitted 2023-09-04; First posted 2023-09-18 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Arm CADe (Active Comparator): Standard, high-definition colonoscopy with the use of CADe assistance (GI-GENIUS, Medtronic; CAD-EYE, Fujifilm; WISE VISION ,NEC). All detected polyps regardless of size and optical diagnosis will be resected and sent to pathology.
  Interventions: Device: Standard, high-definition colonoscopy with the use of CADe assistance
- Standard Arm CADe/CADx (Active Comparator): Standard, high-definition colonoscopy with the use of CADe/CADx assistance (GI-GENIUS, Medtronic; CAD-EYE, Fujifilm; WISE VISION ,NEC). All detected polyps regardless of size and optical diagnosis will be resected and sent to pathology.
  Interventions: Device: Standard, high-definition colonoscopy with the use of CADe/CADx assistance, no leave-in-situ
- Leave-In-Situ Arm (Experimental): Standard, high-definition colonoscopy with the use of CADe/CADx assistance (GI-GENIUS, Medtronic; CAD-EYE, Fujifilm; WISE VISION, NEC).
  Polyps will be left in situ if diminutive (≤5 mm) in size, located in the rectum or sigma and optically diagnosed by the endoscopist using the system to be hyperplastic with high confidence, otherwise resected and sent to pathology.
  Interventions: Device: Standard, high-definition colonoscopy with the use of CADe/CADx assistance, leave-in-situ

INTERVENTIONS:
Device: Standard, high-definition colonoscopy with the use of CADe assistance — All detected polyps regardless of size and optical diagnosis will be resected and sent to pathology.
  Arms: Standard Arm CADe
Device: Standard, high-definition colonoscopy with the use of CADe/CADx assistance, no leave-in-situ — All detected polyps regardless of size and optical diagnosis will be resected and sent to pathology.
  Arms: Standard Arm CADe/CADx
Device: Standard, high-definition colonoscopy with the use of CADe/CADx assistance, leave-in-situ — Polyps will be left in situ if diminutive (≤5 mm) in size, located in the rectum or sigma and optically diagnosed by the endoscopist using the system to be hyperplastic with high confidence, otherwise resected and sent to pathology.
  Arms: Leave-In-Situ Arm

SUMMARY:
This three parallel-arms, randomized, multicenter trial is aimed at investigating the value of AI-assisted optical biopsy for differentiating between neoplastic and non-neoplastic polyps which will lead to the implementation of cost-saving strategies in screening programs. A cost-effectiveness analyses with the use of modern trial emulation analyses of large observational and clinical trial datasets and real-cost data will be conducted. To improve personalized treatment with a novel colonoscopy CADx risk-prediction tool, the investigators will even develop a novel deep learning algorithm for the optical biopsy of the alternative pathway of colorectal cancer carcinogenesis, namely the serrated pathway and develop cost-effectiveness models of AI-assisted optical biopsy in colorectal cancer screening that provides reliable information to identify cancer risk regardless of physicians' skill.

ELIGIBILITY:
Inclusion Criteria:

* All >40 years-old patients undergoing colonoscopy for selected indications

Exclusion Criteria:

* patients with personal history of CRC, or IBD
* patients affected with Lynch syndrome or Familiar Adenomatous Polyposis.
* patients with inadequate bowel preparation (defined as Boston Bowel Preparation Scale <2 in any colonic segment).
* patients with previous colonic resection.
* patients on antithrombotic therapy, precluding polyp resection.
* patients who were not able or refused to give informed written consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority in Adenoma Detection Rate | 4 years
  Non-inferiority in the Adenoma Detection Rate, defined as the proportion of participants with at least one adenoma (per-patient analysis) in the three arms, when adopting a cost-saving leave-in-situ strategy for non-neoplastic rectosigmoid diminutive polyps.

SECONDARY OUTCOMES:
Negative Predictive Value for colorectal neoplasia | 4 years
  Negative Predictive Value for colorectal neoplasia when adopting a leave-in-situ strategy for rectosigmoid diminutive polyps based on the use of Artificial Intelligence.
Concordance between post-polypectomy surveillance and when adopting a leave-in-situ strategy | 4 years
  Concordance between post-polypectomy surveillance based on strategies based on optical diagnosis with Artificial Intelligence and those based on histology, and when adopting a leave-in-situ strategy for colorectal diminutive polyps based on the use of Artificial Intelligence
Change in the cost of polypectomy and histology in screening programs | 4 years
  Change in the cost of polypectomy and histology in screening programs, when implementing strategies based on Artificial Intelligence-based optical biopsy, without changes in benefit related with detection of colorectal neoplasia

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy